CLINICAL TRIAL: NCT01101724
Title: Effect of Early Rest on Recovery From Pediatric Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Danny Thomas, Assistant Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5520163IRC
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Mild Traumatic Brain Injury; Concussion; Post-concussive Syndrome
Keywords: mild traumatic brain injury; Concussion; postconcussive syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): In this group, the treating attending physician will be free to make rest recommendations as they see fit. An internal survey of physician practice found that the vast majority of physicians instruct patients rest for 1-2 days, then to return to school and physical activity after the patient's symptoms have resolved. The amount of rest will vary from patients to patient based on variation in symptom resolution and patient compliance. This advice is consistent with best practices outlined by the CDC.
- Intervention (Experimental): Mandated Rest.
  Interventions: Behavioral: Mandated Rest, Intervention

INTERVENTIONS:
Behavioral: Mandated Rest, Intervention — In addition to CDC based discharge instructions, the intervention group will receive instructions with strict activity restriction explicitly stating "No return to school" and "No Physical Activity" for the next five days. Patients and parents in the intervention group will be provided school and work excuses for the five days post-injury.
  Arms: Intervention

SUMMARY:
The purpose of this study is to find out if strict rest for 5 days helps children get better after concussion.

DETAILED DESCRIPTION:
The purpose of this study is to find out if strict rest for 5 days helps children get better after concussion. This research is being done because, currently, there is no effective treatment for concussion. Physical activity (for example; running, playing sports) and brain activity (for example; homework and tests) may make concussion symptoms worse. We are studying whether strict rest after concussion may help improve symptoms. About 110 children, ages 11-22 years old will take part in this study at the Children's Hospital of Wisconsin. This study is being funded by the Injury Research Center. The research grant pays for study procedures, follow-up testing, and patient reimbursement. Research staff is not being provided incentives to enroll subjects.

ELIGIBILITY:
Inclusion Criteria:

* 11-22 years
* present to the Emergency Department within 24 hours of a head injury

Exclusion Criteria:

* patients who are being admitted,
* non-English speaking patient/family,
* mental retardation (IQ < 70)
* Suspected intoxication
* restricted used of dominant hand or limited vision
* injury or conditions affecting balance assessment
* prior mental defect or disease (e.g., developmental delay, learning disability, or moderate to severe cerebral palsy)
* known intracranial injury (e.g., intracranial bleeding, cerebral contusion)
* patients for whom a legal guardian is not present or cannot be contacted.
* ED clinician preference

Ages: 11 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Outcomes | 10 days post injury
  Neurocogntive outcomes assessed using computer-based neurocogntive testing based on changes from scores obtained in the emergency department to scores obtained at 3 days and 10 days.

SECONDARY OUTCOMES:
Ancillary Neurocogntive Test Battery | 10 days
  Assess neurocognitive outcome using a battery of neuro psych tests at 3 days and 10 days
Parental Attitude to Concussion: | 10 days
  Assess potential barriers to compliance, we will assess parental attitudes toward concussion by administering a survey to parents or caregivers during the ten day home visit.

CONTACTS AND LOCATIONS:
Overall Officials: Danny G Thomas, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Sufrinko AM, Kontos AP, Apps JN, McCrea M, Hickey RW, Collins MW, Thomas DG. The Effectiveness of Prescribed Rest Depends on Initial Presentation After Concussion. J Pediatr. 2017 Jun;185:167-172. doi: 10.1016/j.jpeds.2017.02.072. Epub 2017 Mar 29. PMID 28365025
- [Derived] Silverberg ND, Iverson GL, McCrea M, Apps JN, Hammeke TA, Thomas DG. Activity-Related Symptom Exacerbations After Pediatric Concussion. JAMA Pediatr. 2016 Oct 1;170(10):946-953. doi: 10.1001/jamapediatrics.2016.1187. PMID 27479847
- [Derived] Thomas DG, Apps JN, Hoffmann RG, McCrea M, Hammeke T. Benefits of strict rest after acute concussion: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):213-23. doi: 10.1542/peds.2014-0966. Epub 2015 Jan 5. PMID 25560444